CLINICAL TRIAL: NCT07347392
Title: The Role of Radiotherapy for the Management of Non-melanoma Skin Cancer in Denmark
Acronym: DOSCA-2
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other); Vejle Hospital (Other); Rigshospitalet, Denmark (Other); Copenhagen University Hospital at Herlev (Other); Danish Cancer Society (Other)
Responsible Party: Sponsor
Other Study IDs: DOSCA-2-AUH
Record Dates: First submitted 2025-12-15; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Non-Melanoma Skin Cancer (NMSC); Basal Cell Carcinoma of Skin; Squamous Cell Carcinoma of the Skin
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — Aftercare

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Follow-up visit at least two years after treatment — In Denmark, people treated with primary radiotherapy for NMSC are not routinely offered a hospital follow-up visit to evaluate cosmetic results or recurrence. In this study, patients who received radiotherapy between 2020 and 2024 at five Danish cancer centers will be invited for a clinical examination at least two years after treatment. Cosmetic outcome will be rated by both the patient and a health professional, and any local recurrences will be identified through national health registries.

SUMMARY:
The goal of this observational study is to learn about the long-term effects of radiotherapy for people who were treated for non-melanoma skin cancer (NMSC) in the head and neck area. The study focuses on adults who finished radiotherapy at least two years ago.

The main questions we aim to answer are:

How satisfied are participants with the cosmetic result of their treatment?

What skin changes do healthcare professionals observe at the treated area?

How many participants have experienced a recurrence or developed a new skin cancer, since treatment?

Participants will be invited to:

Attend one extra hospital visit at least two years after they finished radiotherapy

Answer a short questionnaire about their cosmetic satisfaction

Have their skin examined, including photos and dermatoscopy

The results may help improve future treatment guidelines for people with non-melanoma skin cancer.professional, and any local recurrences will be identified through national health registries.

This nationwide study (DOSCA-2) will provide real-world data to help guide future treatment recommendations for NMSC.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Received primary radiotherapy for malignant non-melanoma skin cancer (basal cell carcinoma or cutaneous squamous cell carcinoma) of the head and neck region between 2020 and 2024
* Able to understand and communicate in written and spoken Danish or English

Exclusion Criteria:

* Individuals who are incapable of giving informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults aged 18 years or older with head and neck non-melanoma skin cancer (basal cell carcinoma or cutaneous squamous cell carcinoma) who received primary radiotherapy between 2020 and 2024 at five Danish oncology centres. Participants will be invited via the national digital mailbox (e-Boks) to attend a hospital follow-up visit at the centre where they received radiotherapy, at least two years after completion of treatment. The study represents a real-world national cohort within the Danish public health-care system.
Sampling Method: Non-Probability Sample
Enrollment: 2900 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Cosmetic outcome | At least 2 years after completion of primary radiotherapy for NMSC
  The primary outcome is cosmetic outcome, assessed by both the patient and a health professional using the LENT-SOMA criteria.
Local recurrence | At least 2 years after completion of primary radiotherapy for NMSC
  Identified through the Danish Pathology Registry and follow-up visit

SECONDARY OUTCOMES:
Effect of Tumour Histology | At least 2 years after completion of radiotherapy
  Differences in risk of recurrence between basal cell carcinoma (BCC) and squamous cell carcinoma (SCC) will be analyzed.
Comparison between Short-Course and Long-Course Radiotherapy Regimens | At least 2 years after completion of radiotherapy
  Differences in risk of recurrence between the treatment regimens will be analyzed.
Effect of Tumour Histology | At least 2 years after completion of radiotherapy
  Differences in cosmetic outcome between basal cell carcinoma (BCC) and squamous cell carcinoma (SCC) will be analyzed
Comparison between Short-Course and Long-Course Radiotherapy Regimens | At least 2 years after completion of radiotherapy.
  Differences in cosmetic outcome between the treatment regimens will be analyzed.

OTHER OUTCOMES:
Effect of Treatment-Related Factors | At least 2 years after completion of radiotherapy
  Associations betweem outcomes and field size, field location
Effect of Tumour Related Factors | At least 2 years after completion of radiotherapy
  Associations between outcomes and tumour related factors such as location and TNM stage .
Effect of Patient-Related Factors | At least 2 years after completion of radiotherapy
  Associations between outcomes and patients factors such as age, sex, smoking status, performance status, previous NMSC
Effect of Radiotherapy Modality | At least 2 years after completion of primary radiotherapy for NMSC
  Associations on recurrence and cosmetic outcome depending on radiotherapy modality (kilovoltage (kV), electrons, photons)

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Grau Eriksen, Professor MD PhD, Study Chair — Department of Experimential Clinical Oncology, Aarhus University Hospital, Denmark; Anita Gothelf, MD PhD, Principal Investigator — Department of Oncology, Copenhagen University Hospital, Rigshospitalet, Denmark; Pernille Lassen, MD PhD, Principal Investigator — Department of Oncology, Copenhagen University Hospital, Herlev, Denmark; Rasmus Kjeldsen, MD, Principal Investigator — Department of Oncology, Aalborg University Hospital, Denmark; Gulalai Hanan, MD, Principal Investigator — Department of Oncology, Vejle Hospital, Denmark
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be publicly available due to Danish data protection regulations. Aggregate results will be published in peer-reviewed journals.

REFERENCES:
- [Background] Lansbury L, Leonardi-Bee J, Perkins W, Goodacre T, Tweed JA, Bath-Hextall FJ. Interventions for non-metastatic squamous cell carcinoma of the skin. Cochrane Database Syst Rev. 2010 Apr 14;2010(4):CD007869. doi: 10.1002/14651858.CD007869.pub2. PMID 20393962
- [Background] Thomson J, Hogan S, Leonardi-Bee J, Williams HC, Bath-Hextall FJ. Interventions for basal cell carcinoma of the skin. Cochrane Database Syst Rev. 2020 Nov 17;11(11):CD003412. doi: 10.1002/14651858.CD003412.pub3. PMID 33202063
- [Background] Drucker AM, Adam GP, Rofeberg V, Gazula A, Smith B, Moustafa F, Weinstock MA, Trikalinos TA. Treatments of Primary Basal Cell Carcinoma of the Skin: A Systematic Review and Network Meta-analysis. Ann Intern Med. 2018 Oct 2;169(7):456-466. doi: 10.7326/M18-0678. Epub 2018 Sep 18. PMID 30242379
- [Background] Likhacheva A, Awan M, Barker CA, Bhatnagar A, Bradfield L, Brady MS, Buzurovic I, Geiger JL, Parvathaneni U, Zaky S, Devlin PM. Definitive and Postoperative Radiation Therapy for Basal and Squamous Cell Cancers of the Skin: Executive Summary of an American Society for Radiation Oncology Clinical Practice Guideline. Pract Radiat Oncol. 2020 Jan-Feb;10(1):8-20. doi: 10.1016/j.prro.2019.10.014. Epub 2019 Dec 9. PMID 31831330
- [Background] Zaorsky NG, Lee CT, Zhang E, Keith SW, Galloway TJ. Hypofractionated radiation therapy for basal and squamous cell skin cancer: A meta-analysis. Radiother Oncol. 2017 Oct;125(1):13-20. doi: 10.1016/j.radonc.2017.08.011. Epub 2017 Aug 23. PMID 28843727
- [Background] Schulte KW, Lippold A, Auras C, Bramkamp G, Breitkopf C, Elsmann HJ, Habenicht EM, Jasnoch V, Muller-Pannes H, Rupprecht R, Suter L. Soft x-ray therapy for cutaneous basal cell and squamous cell carcinomas. J Am Acad Dermatol. 2005 Dec;53(6):993-1001. doi: 10.1016/j.jaad.2005.07.045. PMID 16310060
- [Background] Cognetta AB, Howard BM, Heaton HP, Stoddard ER, Hong HG, Green WH. Superficial x-ray in the treatment of basal and squamous cell carcinomas: a viable option in select patients. J Am Acad Dermatol. 2012 Dec;67(6):1235-41. doi: 10.1016/j.jaad.2012.06.001. Epub 2012 Jul 19. PMID 22818756
- [Background] Benkhaled S, Van Gestel D, Gomes da Silveira Cauduro C, Palumbo S, Del Marmol V, Desmet A. The State of the Art of Radiotherapy for Non-melanoma Skin Cancer: A Review of the Literature. Front Med (Lausanne). 2022 Jun 27;9:913269. doi: 10.3389/fmed.2022.913269. eCollection 2022. PMID 35833108
- [Result] Braendstrup ON, Lassen P, Gothelf AB, De Blanck SR, Friborg J, Lonkvist CK, Nielsen AL, Primdahl H, Hanan G, Toure M, Andersen M, Nowicka-Matus K, Kjeldsen R, Eriksen JG. Initial cosmetic outcome six months after kilovoltage therapy of facial basal cell carcinoma: A Danish national prospective study of 932 patients. Sci Rep. 2025 May 29;15(1):18790. doi: 10.1038/s41598-025-03566-8. PMID 40442261
- See also: Cancer Council Australia Keratinoyte Cancer Guidelines Working Party. Clinical Practice Guidelines for Keratinoyte Cancer. 25 Novembe — https://www.cancer.org.au/clinical-guidelines/skin-cancer/keratinocyte-cancer